CLINICAL TRIAL: NCT06350110
Title: T-cell Infusion Targeting BCMA and CD19 for Refractory/Relapsed Systemic Lupus Erythematosus (SLE) Patients With or Without Organs Involvement
Brief Title: Fourth-gen CAR T Cells Targeting BCMA/CD19 for Refractory Systemic Lupus Erythematosus (SLE)
Acronym: BAH242
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202492
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis; Autoimmune Diseases; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatous Polyangiitis; Microscopic Polyangiitis; Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Sjogren's Syndrome
Keywords: CAR-T Cell Therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Autoimmune Diseases; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Scleroderma, Systemic; Myositis; Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
  Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Prior to the infusion of CD19 and BCMA CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for the CAR-T cell therapy to effectively target and eliminate malignant B cells. Following chemotherapy, participants will receive the infusion of CD19 and BCMA CAR-T cells.
  Monitoring and Follow-up:
  Following the CAR-T cell infusion, patients will be subjected to rigorous monitoring to assess safety and treatment response.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Treatment (CD19/BCMA-CAR T cells, chemotherapy) (Experimental): Treatment (CD19/BCMA-CAR T cells, chemotherapy)
  Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive CD19/BCMA-CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of CD19/BCMA-CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of CD19/BCMA-CAR T cells.
  Interventions: Biological: CD19- BCMA CAR-T cells

INTERVENTIONS:
Biological: CD19- BCMA CAR-T cells — The intervention in this clinical trial involves a novel approach using CD19/BCMA-Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  CD19/BCMA-Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, CD19/BCMA-CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial CD19/BCMA-CAR T cell infusion without unacceptable side effects and sufficient CAR T cell availability may receive 2 or 3 additional doses.
  Other Names: EB-BH2024-2

SUMMARY:
This study is a preliminary investigation, with a single-group design, not randomized and transparent, focusing on treatment. Its purpose is to identify the highest dose of BH002 injection (CD19-BCMA CAR-T cells) that patients suffering from resistant systemic lupus erythematosus can tolerate.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a type of autoimmune disorder characterized by the creation of autoantibody-generating immune complexes, affecting various systems and organs.

In SLE, autoreactive B cells can self-activate and morph into plasma cells that produce a high volume of autoantibodies. These cells can also expose their own antigens to autoimmune T cells, thereby stimulating T cells and leading to the release of inflammatory substances.

Conventional treatment for SLE focuses on achieving prolonged remission. In contrast, CD19-BCMA CAR-T cells offer a potential solution by eradicating the abnormal B cells responsible for antibody production. This allows for the rebuilding of the immune system and the restoration of normal immune function in patients, potentially leading to a life free from medication. This highlights the promising potential of CAR-T therapy in treating SLE.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old;
* Total score ≥ 10 on the EULAR/ACR 2019 SLE classification criteria.
* SELENA-SLEDAI≥8.
* Patients with CD19+ B-cell.
* Hemoglobin≥85 g/L.
* WBC≥2.5×10^9/L.
* NEUT≥1×10^9/L.
* BPC≥50×10^9/L.
* AST/ALT below 2 times the upper limit of normal; Creatinine clearance ≥30 mL/min; blood bilirubin ≤2.0 mg/dl; echocardiography indicates that the ejection fraction is ≥50%.
* Adequate venous access for apheresis, and no other contraindications for leukapheresis.
* Women of childbearing age should have a negative serum or urine pregnancy test at screening and baseline.
* Subjects agree to take effective contraceptive measures during the trial until at least 1 year after CAR-T cells infusion.
* Agree to attend follow-up visits as required.
* Voluntary participation and informed consent signed by the patient or his/her legal/authorized representative.

Exclusion Criteria:

* Renal disease: severe lupus nephritis (serum creatinine > 2.5 mg/dL or 221 μmol/L) within 8 weeks --Prior to leukapheresis, or subjects who need hemodialysis.
* CNS disease: including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident [CVA], encephalitis or CNS vasculitis, psychiatric patients with depression or suicidal thoughts.
* Patients with serious lesions and a history of present illness of vital organs such as the heart, liver,kidney blood and endocrine system.
* Patients with immunodeficiency, uncontrolled active infections and active or recurrent peptic ulcers;
* Received immunosuppressive therapy within 1 week prior to leukapheresis.
* Patients with HIV infection; Active infection of hepatitis B virus or hepatitis C virus.
* Patients with syphilis infection.
* The presence or suspicion of an active fungal, bacterial, viral or other infection that cannot be controlled during screening.
* Received live vaccine treatment within 4 weeks prior to screening.
* Severe allergies or hypersensitivity.
* Contraindication to cyclophosphamide in combination with fludarabine.
* Subjects who have undergone major surgery within 2 weeks prior to signing the informed consent form, or who are scheduled to have surgery (other than local anesthetic surgery) during the trial or within 2 weeks of the infusion.
* Cannula or drainage tubes other than central venous catheters.
* Pregnant or lactating women, or subjects who plan to have children within 1 year of treatment;
* Subjects with prior CD19 or BCMA-targeted therapy.
* Participated in any clinical study within 3 months prior to enrollment.
* Subjects with malignant tumour, except for Non-melanoma Skin Cancer with PFS>5yr; Cervical Cancer in situ; Bladder Cancer; Breast Cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/BCMA chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the CD19/BCMA chimeric antigen receptor (CAR) T cells | 10-14 days after apheresis or thawing of cryopreserved peripheral blood mononuclear cell
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No